CLINICAL TRIAL: NCT00369538
Title: Specific Blockage of Angiotensine 2 and Podocyturia in Glomerular Nephropathies With Hypertension and Proteinuria
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: principle investigator moved, new investigators will join, insurance expired - project needs to be re-examined by an ethic committee
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Emmanuel LAVOUE, Directeur Adjoint de la Recherche Clinique et de l'Innovation, University Hospital, Strasbourg, Fance
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3742
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Proteinuria; Hypertension; End Stage Renal Disease
Keywords: Podocyte - podocyturia - microparticles - angiotensin receptor antagonist - glomerulosclerosis; Patients presenting with stable glomerular nephropathy with proteinuria, normal or slightly altered renal function, with hypertension
MeSH Terms: conditions — Proteinuria; Hypertension; Kidney Failure, Chronic | interventions — hydrochlorothiazide, losartan drug combination

ARMS (2):
- 1 (Active Comparator): losartan, hydrochlorothiazide
  Interventions: Drug: losartan, hydrochlorothiazide
- 2 (Active Comparator): hydrochlorothiazide, losartan
  Interventions: Drug: hydrochlorothiazide, losartan

INTERVENTIONS:
Drug: losartan, hydrochlorothiazide — Two administrations of losartan per day,up to 100mg per day, during 2 months, followed by a wash-out during 1 month, and then one administration of hydrochlorothiazide, 25 mg per day during 2 months
  Arms: 1
Drug: hydrochlorothiazide, losartan — One administration of hydrochlorothiazide, 25 mg per day during 2 months, followed by a wash-out during 1 month, and then, two administrations of losartan per day,up to 100mg per day, during 2 months
  Arms: 2

SUMMARY:
Chronic glomerular diseases are one of the main causes leading to end stage renal disease (ESRD). Hypertension and proteinuria are two modifiable factors promoting the progression of ESRD. Podocyte are terminally differentiated epithelial cells and play a central role in the progression of chronic kidney disease and in the development of glomerulosclerosis. The presence of podocyte in urines (podocyturia) has been documented by several teams with continuous and regular podocyturia during glomerular disease. This facts suggests that podocyturia could become a marker of podocyte loss and glomerular damage. In our university hospital, we developed a technique to evaluate the number of microparticles (cellular fragments) in different biologic samples. The podocytary origin of microparticles will be determinated thanks to specific antibodies. The aim of the present study is: i) to quantify podocyturia during glomerular nephropathies by dosing podocyte microparticles ii) to study the relationship between podocyturia and other biologic markers such as proteinuria iii) to evaluate the effect of angiotensine 2 blockage on podocyturia. This is an open-labelled randomized monocenter cross-over study. Twenty subjects with hypertension and glomerular nephropathy characterized by proteinuria and a normal or slightly altered renal function will be included. Patients will be treated successively by an angiotensin receptor blocker (ARB), losartan and by a thiazide, hydrochlorothiazide, (after a wash out period). We will study the impact of these two therapies on podocyturia. Results will be compared with others markers like proteinuria (and its selectivity). We may finally dispose of a non invasive urinary marker of podocyte lesions responsible for glomerulosclerosis and for ESRD progression. Moreover mechanism of nephroprotection of the ARB may be more comprehensive.

ELIGIBILITY:
* Hypertension (TAs > 130, TAd > 80mmHg or under antihypertensive treatment)
* Glomerular nephropathy, proteinuria > 1 g/day, serum creatinin < 200 µmol/L ;
* Informed consent given ;
* No contraindication for ARB and hydrochlorothiazide ;
* Efficient contraception for women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Podocyturia

SECONDARY OUTCOMES:
Proteinuria;
selectivity index of proteinuria
arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Luc FRANTZEN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Néphrologie, Hôpital Civil, Hôpitaux Universitaires, Strasbourg, France